CLINICAL TRIAL: NCT00785486
Title: A Pharmacokinetic Interaction Study Evaluating the Effect of Qualaquin (Quinine Sulfate) Capsules on Midazolam
Brief Title: Drug-Drug Interaction Study of Qualaquin and Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-001-07-1001
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Results first posted 2009-07-08 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: midazolam; drug interactions; cytochrome p450
MeSH Terms: interventions — Midazolam; Quinine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Midazolam alone (Other): Baseline midazolam and 1-hydroxy-midazolam pharmacokinetics. One day 1 after a fast of at least 10 hours patients received a single oral dose of midazolam 2 mg. Blood was drawn at times sufficient to characterize the pharmacokinetics of midazolam and its main metabolite.
  Interventions: Drug: Midazolam Alone
- Qualaquin (quinine) alone steady state (Other): On the morning of day 9 after taking Qualaquin (quinine) capsules 324 mg orally every 8 hours for the prior 5 days, and following a fast of at least 10 hours all study participants received their usual morning dose of Qualaquin (quinine) 324 mg. Blood was drawn at times sufficient to determine the steady state Cmax and AUC 0-tau for Qualaquin (quinine).
  Interventions: Drug: Qualaquin (quinine) alone steady state
- Midazolam with Qualaquin (quinine) (Experimental): On day 10 after taking Qualaquin (quinine) for 6 days according to the stated regimen, all participants took their usual dose of Qualaquin (quinine) with an oral dose of midazolam 2 mg. Blood was drawn sufficient to characterize the steady state kinetics of quinine and the kinetics of midazolam and 1-hydroxy-midazolam in the presence of each other.
  Interventions: Drug: Midazolam and Qualaquin at steady state

INTERVENTIONS:
Drug: Midazolam Alone — Midazolam 2 mg syrup was given orally after a fast of at least 10 hours.
  Other Names: Midazolam
  Arms: Midazolam alone
Drug: Qualaquin (quinine) alone steady state — Qualaquin (quinine) 324 mg capsules were given orally every 8 hours for 7 days ( 21 doses total). On day 9 after taking Qualaquin (quinine) for 5 days according to the stated regimen and fasting for at least 10 hours, all participants took their usual dose of Qualaquin (quinine). Blood was drawn at times sufficient to characterize the pharmacokinetics of quinine at steady state
  Other Names: Qualaquin, Quinine Sulfate
  Arms: Qualaquin (quinine) alone steady state
Drug: Midazolam and Qualaquin at steady state — On the morning of day 10 after taking Qualaquin (quinine) for 6 days according to the stated regimen (324 mg every 8 hours), all participants took their usual dose of Qualaquin (quinine) with an oral dose of midazolam 2 mg after a fast of at least 10 hours
  Other Names: midazolam, Qualaquin, quinine sulfate
  Arms: Midazolam with Qualaquin (quinine)

SUMMARY:
This is an open label non-randomized single sequence, single group two way drug interaction study in healthy adult volunteers to determine the extent to which quinine, an inducer of cytochrome p450 CYP 3A4, affects the pharmacokinetics of midazolam, an accepted probe drug for CYP 3A4. The study will also determine the extent to which midazolam affects the pharmacokinetics of quinine.

DETAILED DESCRIPTION:
This is an open label single sequence single group non-randomized two way drug interaction study in healthy adult volunteers to determine the extent to which quinine, an inducer of cytochrome p450 CYP 3A4, affects the pharmacokinetics of midazolam, an accepted probe drug for CYP 3A4. The study will also determine the extent to which midazolam affects the pharmacokinetics of quinine. This will compare the pharmacokinetics of midazolam and quinine at baseline to their kinetics when they are taken together in 24 normal healthy adult volunteers who will serve as their own controls. All patients will be confined to the study site throughout the entire 11 day study period. On day 1 after a fast of at least 10 hours, all study participants will receive a single oral dose of midazolam 2 mg. Blood will be drawn at times sufficient to adequately define the baseline concentration time curve for midazolam and its metabolite, 1-hydroxy-midazolam. On the morning of day 4, after a 3 day washout period and following a fast of at least 10 hours, all volunteers will begin a regimen of 324 mg of quinine sulfate by mouth every 8 hours. All subjects will continue this regimen from day 4-10 (21 total doses). Blood will be drawn after the first daily dose of quinine on days 4 and 9 at times sufficient to adequately define the baseline and steady state concentration time curves for quinine. Additional blood will be drawn prior to the first daily dose of quinine on days 7,8,9,and 10. On day 10 after a fast of at least a 10 hours, all participants will receive both midazolam 2 mg and quinine 324 mg together. Blood will be drawn a times sufficient to characterize the pharmacokinetics of midazolam, 1-hydroxy-midazolam and quinine under the stated conditions.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy non-smoking, non-obese (≥ 60 kg males, ≥52 kg females within 15% of IBW) adult volunteers 18-45 years of age

Exclusion Criteria:

* Subjects with history or presence of significant cardiovascular disease (including hypotension, hypertension, bradycardia or EKG abnormalities), pulmonary, hepatic, gallbladder or biliary tract, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychiatric disease or an active sexually transmitted disease.
* Subjects with significant blood loss in the prior 56 days, plasma donation within 7 days , hemoglobin < 12.0 g/dl or who have participated in another clinical trial within the prior 30 days.
* Subjects with recent (2-year) history or evidence of alcoholism or drug abuse.
* Subjects who have used any drugs or substances known to inhibit or induce cytochrome P450 (CYP) enzymes 10 days or 28 days respectively prior to the first dose and throughout the study.
* Subjects who have received monoamine oxidase inhibitors or been on a special diet within 28 days of starting the study.
* Subjects who test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV).

Subjects who are pregnant or lactating, taking hormone replacement therapy or have known allergies to quinine sulfate, mefloquine, quinidine or midazolam and other benzodiazepines.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-03; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Davis, MD, Study Chair — Mutual Pharmaceutical; Dennis Swearingen, MD, Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Terkeltaub RA, Furst DE, Digiacinto JL, Kook KA, Davis MW. Novel evidence-based colchicine dose-reduction algorithm to predict and prevent colchicine toxicity in the presence of cytochrome P450 3A4/P-glycoprotein inhibitors. Arthritis Rheum. 2011 Aug;63(8):2226-37. doi: 10.1002/art.30389. PMID 21480191
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Qualaquin (Quinine) And Midazolam Alone And In Combination: All pharmacokinetic studies were begun after a fast of at least 10 hours. On day 1 all participants received a single oral dose of midazolam 2 mg. Blood was drawn at times sufficient to define the baseline kinetics of midazolam and 1-hydroxy-midazolam. After a 3 day washout period, on the morning of day 4, all participants began a regimen of 324 mg of quinine sulfate orally every 8 hours for a total of 21 doses. On day 9 after taking Qualaquin (quinine) for 5 days according to the stated regimen all participants took their usual dose of Qualaquin (quinine). Blood was drawn sufficient to characterize the steady state kinetics of quinine. On day 10 after taking Qualaquin (quinine) for 6 days according to the stated regimen, all participants took their usual dose of Qualaquin (quinine) with an oral dose of midazolam 2 mg. Blood was drawn sufficient to characterize the steady state kinetics of quinine and the kinetics of midazolam and 1-hydroxy-midazolam in the presence of each other.
Period: Midazolam Alone
Arm/Group | Qualaquin (Quinine) And Midazolam Alone And In Combination
Started | 24
Completed | 23 (one participant withdrew for personal reasons after first midazolam dose)
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: 3 Day Washout
Arm/Group | Qualaquin (Quinine) And Midazolam Alone And In Combination
Started | 23
Completed | 23
Not Completed | 0
Period: Qualaquin Alone at Steady State
Arm/Group | Qualaquin (Quinine) And Midazolam Alone And In Combination
Started | 23
Completed | 23
Not Completed | 0
Period: Midazolam With Qualaquin at Steady State
Arm/Group | Qualaquin (Quinine) And Midazolam Alone And In Combination
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Qualaquin (Quinine) And Midazolam Alone And In Combination
Number analyzed (Participants) | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 31.1 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Serum Concentration (Cmax)
Description: Maximum serum concentration(Cmax)
Time Frame: Day 1 (Midazolam Alone), Day 9 (Qualaquin (quinine) Alone), Day 10 Midazolam with Qualaquin (quinine)
Population: per protocol
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Midazolam - Midazolam Alone: On day 1 after a fast of at least 10 hours all participants received a single oral dose of midazolam 2 mg. Blood was drawn at times 0, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 7.917, 12, 15 and 24 hours to determine the baseline Cmax for midazolam.
- 1-Hydroxy-Midazolam - Midazolam Alone: On day 1 after a fast of at least 10 hours all participants received a single oral dose of midazolam 2 mg. Blood was drawn at times 0, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 7.917, 12, 15 and 24 hours to determine the baseline Cmax for 1-hydroxy-midazolam, the primary metabolite of midazolam
- Quinine - Qualaquin(Quinine) Alone: On the morning of day 9 after taking Qualaquin(quinine)capsules 324 mg orally every 8 hours for the prior 5 days, and following a fast of at least 10 hours all study participants received their usual morning dose of Qualaquin (quinine)324 mg. Blood was drawn at times 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, and 7.917 hours to determine the steady state Cmax for Qualaquin (quinine) at this dose.
- Midazolam - Midazolam With Qualaquin(Quinine): On the morning of day 10, after a fast of at least 10 hours all study participants received an oral dose of both midazolam 2 mg and Qualaquin(quinine)324 mg. Blood was drawn at times 0, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 7.917. 12, 15 and 24 hours to determine Cmax for midazolam in the presence of Qualaquin (qunine)at steady state.
- 1-Hydroxy-Midazolam -Midazolam With Qualaquin(Quinine): On the morning of day 10, after a fast of at least 10 hours all study participants received an oral dose of both midazolam 2 mg and Qualaquin(quinine)324 mg concurrently. On day 1 after a fast of at least 10 hours all participants received a single oral dose of midazolam 2 mg. Blood was drawn at times 0, 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 7.917, 12, 15 and 24 hours to determine the Cmax for 1-hydroxy-midazolam in the presence of Qualaquin (quinine) at steady state.
- Quinine - Qualaquin (Quinine) With Midazolam: On the morning of day 10 after taking Qualaquin (quinine)capsules 324 mg orally every 8 hours for the prior 6 days, and following a fast of at least 10 hours all study participants co-ingested oral dose s of midazolam 2 mg and their usual morning dose of Qualaquin (quinine)324 mg. Blood was drawn at times 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, and 7.917 hours to determine the steady state Cmax for Qualaquin (quinine)in the presence of midazolam.
Arm/Group | Midazolam - Midazolam Alone | 1-Hydroxy-Midazolam - Midazolam Alone | Quinine - Qualaquin(Quinine) Alone | Midazolam - Midazolam With Qualaquin(Quinine) | 1-Hydroxy-Midazolam -Midazolam With Qualaquin(Quinine) | Quinine - Qualaquin (Quinine) With Midazolam
Number analyzed (Participants) | 23 | 23 | 23 | 23 | 23 | 23
ng/ml | 12.0435 (3.53669) | 4.6907 (2.17605) | 4432.4089 (678.36810) | 12.5585 (3.51110) | 4.8605 (1.82141) | 4399.7690 (671.04523)

2. Primary Outcome: Area Under the Concentration Time Curve From Zero to T (AUC 0-t) for Midazolam and 1-hydroxy Midazolam at Baseline and With Qualaquin (Quinine) at Steady State.
Description: Area under the concentration time curve(AUC 0-t) calculated by the linear trapezoidal method from time 0 to 24 hours, for Midazolam and 1-hydroxy-midazolam on day 1 (midazolam alone) and day 10 (midazolam with Qualaquin -(quinine) at steady state to determine if a significant drug interaction occurs between midazolam and quinine
Time Frame: Days 1 and 10 at 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 7.917, 12, 15 and 24 hours
Population: by protocol
Measure: Mean (Standard Deviation); unit: ng•h/mL
Groups:
- Midazolam - Midazolam Alone: On day 1 after a fast of at least 10 hours all participants received a single oral dose of midazolam 2 mg. Blood was drawn at times sufficient to characterize the Area under the concentration time curve from zero to 24 hours (AUC 0-t) of midazolam and 1-hydroxymidazolam
- 1-Hydroxy-Midazolam - Midazolam Alone: On day 1 after a fast of at least 10 hours all partcipants received a single oral dose of midazolam 2 mg. Blood was drawn at times sufficient to characterize the Area under the concentration time curve from zero to 24 hours (AUC 0-t) of 1-hydroxy midazolam as calculated by the linear trapezoidal method.
- Midazolam - Midazolam With Qualaquin (Quinine): On day 10 after a fast of at least 10 hours all partcipants received a single oral dose of midazolam 2 mg and Qualaquin (quinine) 324 mg. Blood was drawn at times sufficient to characterize the Area under the concentration time curve from zero to 24 hours (AUC 0-t) for midazolam in the presence of Qualaquin(quinine)at steady state as calculated by the linear trapezoidal method.
- 1-Hydroxy-Midazolam -Midazolam With Qualaquin (Quinine): On day 10 after a fast of at least 10 hours all partcipants received a single oral dose of midazolam 2 mg and Qualaquin (quinine) 324 mg. Blood was drawn at times sufficient to characterize the Area under the concentration time curve from zero to 24 hours (AUC 0-t) for 1-hydroxy midazolam in the presence of Qualaquin(quinine)at steady state as calculated by the linear trapezoidal method.
Arm/Group | Midazolam - Midazolam Alone | 1-Hydroxy-Midazolam - Midazolam Alone | Midazolam - Midazolam With Qualaquin (Quinine) | 1-Hydroxy-Midazolam -Midazolam With Qualaquin (Quinine)
Number analyzed (Participants) | 23 | 23 | 23 | 23
ng•h/mL | 30.076 (10.1593) | 10.780 (6.6534) | 27.242 (6.5008) | 10.454 (5.2714)

3. Primary Outcome: Area Under the Concentration Time Curve From Zero to Infinity (AUC Inf) for Midazolam and 1 Hydroxy Midazolam Before (Day 1) and After (Day 10) Qualaquin (Quinine).
Description: AUC inf for Midazolam and hydroxy-midazolam on day 1 (midazolam alone) and day 10 (midazolam with steady state Qualaquin(quinine)- the sum of AUC0-t plus the ratio of the last measured plasma concentration to the elimination rate constant to determine whether a significant drug interaction occurs between midazolam and quinine
Time Frame: Days 1 and 10 at 0.167, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 7.917, 12, 15 and 24 hours
Population: per protocol
Measure: Mean (Standard Deviation); unit: ng·h/mL
Groups:
- Midazolam - Midazolam Alone: On day 1 after a fast of at least 10 hours all partcipants received a single oral dose of midazolam 2 mg. Blood was drawn sufficient to characterize AUC inf for midazolam alone calculated as the sum of AUC0-t plus the ratio of the last measurable plasma concentration to the elimination rate constant
- 1-Hydroxy-Midazolam - Midazolam Alone: On day 1 after a fast of at least 10 hours all participants received a single oral dose of midazolam 2 mg. Blood was drawn sufficient to characterize AUC inf for 1-hydroxy-midazolam alone calculated as the sum of AUC0-t plus the ratio of the last measurable plasma concentration to the elimination rate constant.
- Midazolam - Midazolam With Qualaquin (Quinine): On day 10 after a fast of at least 10 hours all partcipants received a single oral dose of midazolam 2 mg and Qualaquin (quinine) 324 mg . Blood was drawn sufficient to characterize AUC inf for midazolam alone calculated as the sum of AUC0-t plus the ratio of the last measurable plasma concentration to the elimination rate constant
- 1-Hydroxy-Midazolam -Midazolam With Qualaquin (Quinine): On day 10 after a fast of at least 10 hours all partcipants received a single oral dose of midazolam 2 mg and Qualaquin(quinine) 324 mg. Blood was drawn sufficient to characterize AUC inf for 1- hydroxy-midazolam alone calculated as the sum of AUC0-t plus the ratio of the last measurable plasma concentration to the elimination rate constant
Arm/Group | Midazolam - Midazolam Alone | 1-Hydroxy-Midazolam - Midazolam Alone | Midazolam - Midazolam With Qualaquin (Quinine) | 1-Hydroxy-Midazolam -Midazolam With Qualaquin (Quinine)
Number analyzed (Participants) | 23 | 23 | 23 | 23
ng·h/mL | 31.324 (10.0930) | 11.669 (7.4340) | 28.771 (6.8081) | 11.447 (5.8587)

4. Primary Outcome: The Area Under the the Concentration Time Curve From Zero to Tau (0-8hrs) for Qualaquin (Quinine) AUC Tau Before and After Midazolam
Description: Qualaquin (quinine) - AUC tau alone at steady state (day 9) and in the presence of coadministered midazolam 2 mg (day 10) over the dosing interval (0 - 8 hours), as calculated by the linear trapezoidal method.
Time Frame: Days 9 and 10 at 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, and 7.917 hours
Population: per protocol
Measure: Mean (Standard Deviation); unit: ng•h/mL
Groups:
- Qualaquin (Quinine) Alone: On the morning of day 9 after taking an oral dose of Qualaquin quinine)324 mg every 8 hours for the prior 5 days (Steady state) and following a fast of at least 10 hours all participants took a an additional 324 mg oral dose of the drug. Blood was drawn sufficient to determine the pharmacokinetics of Qualaquin(Quinine) alone over the following dosing interval (0 - 8 hours), as calculated by the linear trapezoidal method.
- Qualaquin (Quinine) With Midazolam: On day 10 after six days of receiving Qualaquin 324 mg every 8 hours, and after a fast of at least 10 hours, patients received a 2 mg dose of midazolam and 324 mg of Qualaquin (quinine)(Steady state). Blood was drawn sufficient to determine the pharmacokinetics of Qualaquin(quinine) in the presence of midazolam over the final dosing interval (0 - 8 hours), as calculated by the linear trapezoidal method.
Arm/Group | Qualaquin (Quinine) Alone | Qualaquin (Quinine) With Midazolam
Number analyzed (Participants) | 23 | 23
ng•h/mL | 30455.4 (5028.27) | 30568.7 (4851.10)

ADVERSE EVENTS:
Groups:
- Midazolam Alone: Adverse effects on day 1 after participants received 2mg of midazolam syrup orally.
- Qualaquin (Quinine) Alone: Adverse effects(ADR)while taking Qualaquin(quinine)324 mg alone orally every 8 hours on days 4-11. Results are reported as total for the 7 day period.
- Midazolam With Qualaquin (Quinine) Together: Adverse effects reported on day 10 after participants received 2 mg of midazolam syrup and 324 mg of Qualaquin(quinine)orally.
Arm/Group | Midazolam Alone | Qualaquin (Quinine) Alone | Midazolam With Qualaquin (Quinine) Together
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 1 | 27 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 4.3% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Midazolam Alone | Qualaquin (Quinine) Alone | Midazolam With Qualaquin (Quinine) Together
Headache (Nervous system disorders) | 0/23 (0) | 10/23 (10) | 3/23 (3)
Tinnitis (Ear and labyrinth disorders) | 1/23 (1) | 4/23 (4) | 0/23 (0)
Feeling Hot (General disorders) | 0/23 (0) | 4/23 (4) | 0/23 (0)
Nausea (Gastrointestinal disorders) | 0/23 (0) | 3/23 (3) | 1/23 (1)
Tremor (Nervous system disorders) | 0/23 (0) | 3/23 (3) | 0/23 (0)
Ear Discomfort (Ear and labyrinth disorders) | 0/23 (0) | 3/23 (3) | 0/23 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days